CLINICAL TRIAL: NCT06318416
Title: Precision Rifampin (P-RIF) Trial for Personalized Dosing in Active Tuberculosis Disease
Brief Title: Precision Rifampin Trial for Personalized Dosing
Acronym: P-RIF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Rutgers University (Other); Haydom Lutheran Hospital (Other)
Responsible Party: Principal Investigator, Scott Heysell, MD, Associate Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HSR230382
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early (Experimental): Urine spectrophotometry for rifampin absorbance and rifampin dose adjustment at Day 14
  Interventions: Diagnostic Test: urine spectrophotometry for rifampin absorbance
- Delayed (Experimental): Urine spectrophotometry for rifampin absorbance and rifampin dose adjustment at Day 21
  Interventions: Diagnostic Test: urine spectrophotometry for rifampin absorbance

INTERVENTIONS:
Diagnostic Test: urine spectrophotometry for rifampin absorbance — All participants will received conventional weight-based TB therapy, standard of care for active TB disease. After enrollment, participants will be randomized to early Day 14 or delayed Day 21 dose modification of rifampin informed by urine spectrophotometry where absorbance is determined above or below a threshold. Below a threshold, single tablets of rifampin are added to conventional fixed drug combination standard of care, above a threshold, no additional rifampin is added. Dose adjustment of rifampin may be up to ~30mg/kg and will be continued through day-56.

SUMMARY:
Individual pharmacokinetic variability is an important driver of tuberculosis (TB) treatment failure particularly among undernourished populations, and that suboptimal serum drug concentrations are associated with delayed response to treatment, death, and acquired bacterial drug resistance. Serum drug exposures can be approximated by urine excretion as measured by spectrophotometry, replacing the need for specialized equipment for serum testing. Anti-TB pharmacokinetic variability has also been associated with enteric pathogen burden. The overall hypothesis is that urine spectrophotometry will identify people with below-target rifampin serum concentrations, which can be corrected to target levels after dose adjustment as confirmed by serum mass spectrometry. Therefore, this protocol includes a clinical trial to assess efficacy and safety of rifampin dose adjustment based on urinary excretion levels among adults and children who are being treated for drug-sensitive pulmonary TB at our longstanding collaborative research site in Haydom Lutheran Hospital, Tanzania.

DETAILED DESCRIPTION:
This is a single-site trial at Haydom Lutheran Hospital, a regional referral hospital level in Manyara Region of northern Tanzania. The primary objective: Among children and adults in Tanzania initiating treatment for drug-susceptible pulmonary TB, perform urine spectrophotometric testing for rifampin, and collect serum throughout the 24 hour dosing interval for later concentration measurement by gold-standard mass spectrometry and comparative pharmacokinetics. Patients with urine rifampin excretion below target will undergo incremental dose increase and urine spectrophotometry and serum collection will be repeated. Stool will also be evaluated at regular intervals to understand the association with enteropathogen burden and effects on rifampin absorption, urine excretion, and serum exposures. Participants will randomized to an early group where urine spectrophotometry and dose adjustment is performed at Day 14 after treatment initiation, or a delayed group where the intervention is performed at Day 21. Primary efficacy endpoint is the proportion of subjects in the early and delayed groups that reach serum target AUC0-24 (35 ug/mL for adults; 31.7 ug/mL for children) at Day 21, before the urine based dose adjustment is made in the delayed group. Primary safety endpoint is the number of severe adverse events. Secondary endpoints include: time to sputum culture conversion to negative, weight change. Time to culture conversion and weight change are stratified by age given pediatric populations are more likely to be culture negative and clinically diagnosed with weight gain a central measurement of treatment response. Safety of dose adjustment strategy parameters include clinical adverse events, liver function tests, kidney function tests and hematological parameters

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 or older
2. Diagnosed with active, rifampin-susceptible, pulmonary TB- sputum positive for M. tuberculosis complex without rpoB mutation, or culture for M. tuberculosis with conventional rifampin susceptibility OR among children unable to expectorate, meeting confirmed or probable consensus clinical case definitions for intrathoracic childhood TB
3. Initiating combination anti-TB therapy with isoniazid, rifampin, pyrazinamide, and ethambutol
4. Subject or guardian is able to provide informed consent; and for children 7 years or older, provide assent
5. Stated willingness to comply with all trial procedures and availability for the duration of the trial
6. Resident within a pre-defined geographic area to ensure TB clinic follow-up

Exclusion Criteria:

1. Urinary incontinence: may complicate urine collection
2. Oliguria: may complicate urine collection and limit correlation of urinary excretion and serum concentrations
3. Kidney disease, defined as a glomerular filtration rate (GFR) < 60 mL/min: In 5R01 AI137080, those adults with GFR < 60 mL/min had reduced correlation or urinary rifampin excretion and serum concentrations.
4. Severe anemia, defined as a hemoglobin level less than 7 g/dL: given planned phlebotomy
5. Elevated liver function tests, defined as DAIDS grade 3 or above (ALT or AST >/= 5 x upper limit of normal): may confound potential toxicity signals of dose adjustment strategy
6. Pregnancy: Urine rifampin spectrophotometry has not been studied in pregnant people, higher dose rifampin also less studied in pregnancy, and may confound potential toxicity signals (e.g. elevated liver function tests in pregnancy). Urine pregnancy test will be completed at screening in people of child-bearing potential. Child-bearing potential is defined as a person able to menstruate (menstruation in the last 12 months) and not receiving a form of contraception with less than <1% failure rate (oral levonorgestrel, IUD or etonogestrel implant).
7. Weight <10.0 kg (dose increase may exceed 30mg/kg/dose)
8. Current treatment with a drug known to have significant interaction with anti-TB therapy
9. Excessive alcohol use? (for example, Men consuming > 14 standardized drinks per week and/or > 4 drinks per day OR women consuming >7 standardized drinks per week, and/or >3 drinks per day, or at the discretion of the investigator(s).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Rifampin serum area under the concentration time curve for the 24 hour dosing interval | 21 days
  Primary efficacy endpoint is the proportion of subjects in the early and delayed group that reach serum target AUC0-24 (35 ug/mL for adults; 31.7 ug/mL for children).
Adverse events | 56 days
  Primary safety endpoint is the number of serious adverse events

SECONDARY OUTCOMES:
Time to sputum culture conversion to negative | 56 days
  Time to sputum culture conversion to negative from pretreatment, Day 0, and serial sample collection as measured by mycobacterial load assay
Weight change | 56 days
  Percent of weight change of total body weight in kilograms
Enteropathogen burden | 14, 21 and 28 days after enrollment
  Total number of enteropathogen species as detected by stool multiplex PCR TaqMan Array Card
Biomarkers of intestinal inflammation, permeability and intestinal mass | 14, 21, 28 days after enrollment
  Serum citruline, stool myeloperoxidase, stool alpha-1-antitrypsin, stool neopterin

CONTACTS AND LOCATIONS:
Locations (1):
- Haydom Lutheran Hospital, Haydom, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xie YL, Modi N, Handler D, Yu S, Rao P, Kagan L, Petros de Guex K, Reiss R, Siemiatkowska A, Narang A, Narayanan N, Hearn J, Khalil A, Woods P, Young L, Lardizabal A, Subbian S, Peloquin CA, Vinnard C, Thomas TA, Heysell SK. Simplified urine-based method to detect rifampin underexposure in adults with tuberculosis: a prospective diagnostic accuracy study. Antimicrob Agents Chemother. 2023 Nov 15;67(11):e0093223. doi: 10.1128/aac.00932-23. Epub 2023 Oct 25. PMID 37877727
- [Background] Thomas TA, Lukumay S, Yu S, Rao P, Siemiatkowska A, Kagan L, Augustino D, Mejan P, Mosha R, Handler D, Petros de Guex K, Mmbaga B, Pfaeffle H, Reiss R, Peloquin CA, Vinnard C, Mduma E, Xie YL, Heysell SK. Rifampin urinary excretion to predict serum targets in children with tuberculosis: a prospective diagnostic accuracy study. Arch Dis Child. 2023 Aug;108(8):616-621. doi: 10.1136/archdischild-2022-325250. Epub 2023 Apr 25. PMID 37171408